CLINICAL TRIAL: NCT03291925
Title: Primary Non-invasive Cardiac Computed Tomography Versus Routine Invasive Angiography Prior to TAVI: A Randomized Controlled Pilot Trial (CT-CA Study)
Brief Title: Primary Non-invasive Cardiac Computed Tomography Versus Routine Invasive Angiography Prior to TAVI
Acronym: CT-CA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: BC Centre for Improved Cardiovascular Health (Other)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ICVHealth2016002
Record Dates: First submitted 2017-03-28; First posted 2017-09-25 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Severe Aortic Stenosis; Transcatheter Aortic Valve Implantation
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, open-label trial.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Selective invasive angiography based on CT/CCTA imaging (Experimental): Patients will undergo selective invasive angiography based on CT/CCTA imaging. Decision to procede with additional invasive CA will be based on adequacy of CT/CCTA evaluation and likelihood of significant coronary artery disease.
  Interventions: Procedure: Selective invasive angiography based on CT/CCTA imaging.
- Invasive Cardiac Angiography (Active Comparator): Patients will undergo systematic invasive angiography.
  Interventions: Procedure: Procedure/Surgery: Invasive angiography

INTERVENTIONS:
Procedure: Selective invasive angiography based on CT/CCTA imaging.
  Arms: Selective invasive angiography based on CT/CCTA imaging
Procedure: Procedure/Surgery: Invasive angiography
  Arms: Invasive Cardiac Angiography

SUMMARY:
This pilot study is a prospective, randomized, open-label trial that aims to assess the feasibility of comparing a primary Computed tomography/Cardiac computed tomography angiography (CT/CCTA) strategy (test arm) to a strategy combining routine use of CT/CCTA and invasive CA (control arm) prior to a Transcatheter aortic valve implantation (TAVI) procedure. The study will also estimate the rate of composite coronary adverse events (myocardial infarction, post procedural coronary revascularization and cardiovascular mortality) between the two arms at 90 days follow-up. The primary endpoint will be the feasibility of recruitment and compliance with the study protocol at 2 sites in Canada and 1 site in Denmark. Additional clinical endpoints including: all-cause death at 90 days post procedure, myocardial infarction at 90 days post procedure, unplanned PCI or CABG at 90 days post procedure, stroke at 90 days post procedure, CA and PCI related cumulative vascular complications events. This information will be used to inform the design of the definitive efficacy trial.

ELIGIBILITY:
Inclusion Criteria:

* Severe aortic stenosis (Peak transvalvular gradient of ≥ 40mmHg on TTE or stress Echo, Aortic valve area of < 1.0cm2)
* Symptoms suggestive of aortic stenosis (dyspnea, syncope, angina)
* Eligible for TAVI (Upon evaluation by a multidisciplinary team composed of at least one interventional cardiologist and one cardiothoracic surgeon)

Exclusion Criteria:

* Severe renal dysfunction Glomerular filtration rate < 30 ml/min.
* Severe left ventricular dysfunction LVEF ≤ 30%
* Recent coronary angiography ≤ 6months from randomization
* Recent PCI ≤ 6months from randomization
* Recent or active acute coronary syndrome (New or worsening angina with or without positive biomarkers or ECG changes).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-11; Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Number of patients enrolled in the study of all those that are eligible | 18 months
  This is the primary outcome for this pilot study to assess feasibility of a larger trial.

SECONDARY OUTCOMES:
All-cause mortality | 90 days
Myocardial Infarction | Peri-procedural (≤72h post procedure) and 90 days
  According to Valvular Academic Research Consortium-2 (VARC-2) criteria.
  * Periprocedural MI (≤72h post procedure).
  * Spontaneous MI.
Unplanned revascularization | 90 days
  Any unplanned coronary revascularization either with Percutaneous Coronary Intervention( PCI) or Coronary Artery Bypass Graft (CABG) post TAVI procedure.
Bleeding complication | Peri-procedural (≤72h post procedure) and 90 days
  According to VARC-2 criteria.
  * TAVI related ≤ 72h post TAVI
  * Coronary procedure related ≤ 72h post CA or PCI (if staged TAVI-PCI)
Device success | 90 days
  According to VARC-2 criteria.
Acute Kidney Injury | 90 days
  According to VARC-2 criteria.
Stroke | 90 days
  An acute episode of focal or global neurological dysfunction caused by the brain, spinal cord, or retinal vascular injury as assessed by a clinician and confirmed by at least one cerebral imaging study (CT or MRI). Stroke may be classified as ischaemic or haemorrhagic

CONTACTS AND LOCATIONS:
Overall Officials: Jonathon Leipsic, MD, Principal Investigator — St. Paul's Hospital
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No